CLINICAL TRIAL: NCT01560546
Title: Testosterone Therapy of Men With Type 2 Diabetes Mellitus (T2DM) - a Randomised, Doubleblinded and Placebocontrolled Trial of Men With Subnormal Testosterone Levels and T2DM.
Brief Title: Testosterone Therapy of Men With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marianne Andersen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Marianne Andersen, MD, ph.d., Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-002102-73
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes Mellitus; Hypogonadism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testim (Active Comparator)
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Placebo for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — 50 mg/dose/day for 24 weeks
  Other Names: Testim
  Arms: Testim
Drug: Placebo — placebo on the skin for 24 weeks
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled, double-blinded study on 40 men with type 2 DM.

Type 2 diabetes mellitus (T2DM) is a common endocrine disorder characterized by hyperinsulinaemia and insulin resistance.

Hypothesis Testosterone therapy increases lean body mass and insulin sensitivity in men with low normal levels of bioavailable testosterone and type 2 DM.

DETAILED DESCRIPTION:
Background Inadequate levels of androgens have been associated with an increased risk of chronic illnesses including obesity and diabetes. Moreover, testosterone treatment has been shown to increase lean body mass and lipid oxidation as well as insulin sensitivity in hypogonadal men.

ELIGIBILITY:
Inclusion Criteria:

* Male gender age 50-70
* Bioavailable testosterone < 7,3 nmol/L
* Metformin treatment of T2DM for 3 months or more

Exclusion Criteria:

* HbA1c > 9,0 %, BMI > 40 kg/m2, Haematocrit > 50%,
* Known malignant disease, PSA > 3 ug/L, Nycturia > 3 times,
* Abnormal routine blood samples,
* Severe hypertension,
* Significant EKG-changes,
* Wish of parenthood,
* Active mental illness,
* former or present abuse,
* Severe illness of heart-, lung- or kidney,
* Primary or secondary hypogonadism.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Lean body mass | approximately three years
  Accessed by DXA scanning

SECONDARY OUTCOMES:
Insulin sensitivity | three years
  Euglycemic hyperinsulinaemic clamp
Regional body composition and liver fat | three years
  DXA- and MR-scans and spect
Glucose and lipid oxidation | three years
  Indirect calorimetry
Myostatin and satellite cells | 8 years
  Muscle biopsy
Inflammation | 8 years
  Hormones: Adiponectin, leptin osteoprotegerin, IGF-I, bioactive IGF-I, Urine cortisol and steroid metabolites etc.
Physical activity | three years
  Questionaires
Quality of life | three years
  Questionaires
Sexual function | Three years
  Questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, MD, ph.d., Principal Investigator
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Botha J, Velling Magnussen L, Nielsen MH, Nielsen TB, Hojlund K, Andersen MS, Handberg A. Microvesicles Correlated with Components of Metabolic Syndrome in Men with Type 2 Diabetes Mellitus and Lowered Testosterone Levels But Were Unaltered by Testosterone Therapy. J Diabetes Res. 2017;2017:4257875. doi: 10.1155/2017/4257875. Epub 2017 Jan 12. PMID 28168203